CLINICAL TRIAL: NCT06188234
Title: Observational Study on the Prescription Patterns and Clinical Efficacy of Tenero Tab/Tenero M SR Tab in Korean Type 2 Diabetes Mellitus Patients
Brief Title: The Prescription Patterns and Clinical Efficacy of Tenero Tab/Tenero M SR Tab
Status: Recruiting | Type: Observational
Sponsor: Hanlim Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-TNL/M-401
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metformin HCI; Teneligliptin hydrochloride
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to observe the prescription patterns and clinical efficacy of patients prescribed with Tenero Tab/Tenero M SR Tab for diabetes treatment in routine clinical practice.

DETAILED DESCRIPTION:
This study is to observe the clinical efficacy by analyzing the prescription patterns in routine clinical practice and changes in HbA1c, FPG, PP2G, etc., of patients prescribed with Tenero Tab/Tenero M SR Tab for diabetes treatment. Additionally, the study intends to assess patient satisfaction based on these observations.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 19 years of age
2. Individuals diagnosed with type 2 diabetes.
3. Individuals who, at the clinical discretion, are prescribed Tenero Tab or Tenero M SR Tab for the purpose of diabetes treatment for the first time.
4. Individuals who have voluntarily provided written consent to participate in this study.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Individuals who are contraindicated according to the approved indications of Tenero Tab/Tenero M SR Tab.
3. Other cases where the principal investigator and study personnel deem individuals ineligible for participation in this clinical trial.

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients prescribed Tenero Tab/Tenero M SR Tab for diabetes treatment.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c at 6 months of prescribing Tenero Tablet/Tenero Emextended Release Tablet compared to baseline | after 6 months of prescription for Tenero Tab/Tenero M SR Tab compared to baseline
  Change in HbA1c at 6 months of prescribing Tenero Tablet/Tenero Emextended Release Tablet compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Seokgi Yoon, Principal Investigator — CHEONAN ENDO MEDICAL CLINIC
Locations (1):
- Cheonan Endo Medical Clinic, Cheonan, South Korea